CLINICAL TRIAL: NCT01243255
Title: Centralized Pan-European Survey on the Undertreatment of Hypercholesterolemia. Polish Survey on the Efficacy of the Hypercholesterolemia Treatment
Brief Title: Polish Survey on the Efficacy of the Hypercholesterolemia Treatment
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CPL-DUM-2010/1
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; low density lipoprotein; undertreatment of hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with hypercholesterolemia on lipid lowering pharmacological treatment

SUMMARY:
The purpose of the survey is to evaluate the efficacy of treatment of hypercholesterolemia in Polish patients who are currently on lipid- lowering pharmacological therapy . Efficient treatment is defined as achievement of the LDL cholesterol level goals according to the European Society of Cardiology 2007 guidlines.

ELIGIBILITY:
Inclusion Criteria:

* Patients on lipid lowering drug treatment
* Lipid lowering drug treatment lasting at least 3 months
* No lipid lowering drug/dose change for a minimum 6 weeks prior to enrolment to the study

Exclusion Criteria:

* Lack of patient's signed informed consent form
* Lack of the blood sample taken for lipid profile and glucose within 10 days before or after assessment of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
establish the proportion of patients on lipid lowering pharmacological treatment reaching the LDL-C goals according to ESC 2007 guidelines in general. | whole study procedure takes place during the one, single patient's visit

SECONDARY OUTCOMES:
establish the proportion of patients on lipid lowering pharmacological treatment in primary prevention, reaching the LDL-C goals according to ESC 2007 guidelines for this sub-population | whole study procedure takes place during the one, single patient's visit
establish the proportion of patients on lipid lowering pharmacological treatment in secondary prevention, reaching the LDL-C goals according to ESC 2007 guidelines for this sub-population | whole study procedure takes place during the one, single patient's visit
identify determinants (patient and physician characteristics) for undertreatment of hypercholesterolemia. | whole study procedure takes place during the one, single patient's visit

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Artur Mamcarz, Principal Investigator — Medical University of Warsaw; Barbara Możejko-Pastewka, Study Director — AstraZeneca Pharma